CLINICAL TRIAL: NCT03587857
Title: A Mobile Health Application for Engagement in Care Among Youth Living With HIV
Brief Title: mHealth App for Engagement in Care Among Youth Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R34MH114604 (NIH); R34MH114604 (NIH)
Record Dates: First submitted 2018-04-29; First posted 2018-07-16 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: HIV/AIDS; Mobile Health; Young Adults
Keywords: Health Disparity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1: Intervention (Experimental): All YLWH who choose to enroll in the study will receive access to WYZ, the mobile health application. The participants will be asked to use the app for 6 months, during which the investigators will assess the feasibility and acceptability of WYZ. Based on this initial data, the investigators will refine and release a new version of the app (WYZ 3.0).
  Interventions: Other: Mobile Health Application

INTERVENTIONS:
Other: Mobile Health Application — This mobile health app is a modular, adaptive, and personalized intervention delivered via a mobile phone. It is grounded in the Information Motivation Behavioral Skills (IMB) model. It was created in collaboration with YLWH (18-29 years-old) using a Human-Centered Design approach to help improve engagement in HIV care among this age group.
  Other Names: WYZ

SUMMARY:
In the US, fewer than 6% of all youth living with HIV (YLWH) achieve HIV viral suppression. However, health disparities among youth extend across the entire HIV care continuum in that there is a strong association between younger age and later HIV diagnosis, lower engagement in care, lower levels of antiretroviral therapy (ART) adherence, and worse HIV clinical outcomes. In response to this critical public health dilemma, the investigators propose to develop a novel mobile health application ("app") to improve engagement in health care and ART adherence and to pilot test this mobile health app in 18-29-year-old YLWH residing in San Francisco.

The aims of this study are to:

Aim 1: Build on a theory-guided model and formative work to complete the development of a novel personalized mobile health app for improved HIV clinical outcomes among YLWH (includes field test of initial release to ensure adequate usability and engagement).

Aim 2: Conduct a six-month single arm pilot study to examine WYZ feasibility and acceptability among YLWH ( N = 76) living in the San Francisco Bay Area. Finally, the investigators will conduct in-depth qualitative interviews with a subset of participants (N = 20) and clinical team members (N = 10) whose patients participated in the pilot study.

The investigators hypothesize that this mobile health app will be feasible and acceptable and will result in improved HIV clinical outcomes. Upon completion, the investigators will be ready to test the efficacy of this app in a subsequent large-scale randomized control trial among a population that is disproportionately impacted by HIV and at elevated risk for poor clinical outcomes.

DETAILED DESCRIPTION:
WYZ is a modular, adaptive, and personalized intervention delivered via a mobile phone. It is grounded in the Information-Motivation-Behavioral Skills (IMB) model which has been valuable for understanding and guiding the development of interventions for complex health behaviors. WYZ was created in collaboration with 18-29 year-old YLWH using a Human-Centered Design (HCD) approach that emphasizes understanding the perspective of the users of the technology. WYZ is intended to improve engagement in HIV care by 1) enhancing medication adherence self-efficacy, 2) increasing awareness and use of community resources, 3) reducing barriers to communication between youth and their healthcare team, and 4) providing a secure platform for the formation of a supportive closed online community of YLWH.

The investigators will complete development of WYZ (1.0), field test the initial release with a cohort of 10 potential users over a period of three months to identify and address technical challenges, and develop a fully functioning version (WYZ 2.0) that can be used in a pilot investigation. The investigators will then conduct a six-month single-arm pilot study to examine WYZ feasibility and acceptability among (N = 76) YLWH (18-29 years old) who live and/or receive care in the San Francisco Bay Area. The objectives of this forthcoming phase are to refine the design so as to improve satisfaction and engagement with the intervention among YLWH and their healthcare providers.

The main outcomes of the pilot trial include feasibility and acceptability as indicated by meeting or exceeding proposed benchmarks. Feasibility will be assessed via user metrics by examining the participant's interactions with WYZ via a mobile analytics service called Flurry and backend (Salesforce) reporting tools. Acceptability will be examined during regular phone check-ins, a system usability scale (SUS), a satisfaction survey, and an exit qualitative interview.

In addition to feasibility measures, the investigators will calculate an engagement index (EI) for each participant. The EI has been detailed and used successfully in other mHealth interventions. The EI includes the following sub-indices: (1) click depth (number of pages a user views per session), (2) loyalty (measures how frequently users access the application during the study period), (3) recency (the time difference between each session the user accessed the application), (4) interaction (number of push notifications opened from those sent through the application), and (5) feedback (subjective measure of participants' satisfaction with the application).

Based on the data from participants in this pilot study, the investigators will develop a refined version of WYZ (3.0), which will be used in a future investigation to examine the efficacy of the intervention with a much larger sample.

ELIGIBILITY:
Eligibility Criteria:

* Must be between 18 and 29 years of age
* Must be living with HIV
* Must reside and/or get care in San Francisco Bay Area
* Must be able to provide informed consent to be a research participant
* Must be able to speak and understand English
* Must have access to an Android (5.0 or higher) or iOS (10.0 or higher) mobile phone

Exclusion Criteria:

Evidence of cognitive impairment or psychotic disorder that prevents one from understanding the purpose of the study and/or participating fully in study activities. This determination will be made by trained study staff in consultation with the principal investigator.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parya Saberi, PhamD, Principal Investigator — UCSF School of Medicine, Division of Prevention Science
Locations (1):
- University of California San Francisco, Mission Bay Campus, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erguera XA, Johnson MO, Neilands TB, Ruel T, Berrean B, Thomas S, Saberi P. WYZ: a pilot study protocol for designing and developing a mobile health application for engagement in HIV care and medication adherence in youth and young adults living with HIV. BMJ Open. 2019 May 5;9(5):e030473. doi: 10.1136/bmjopen-2019-030473. PMID 31061063
- [Result] Saberi P, Lisha NE, Erguera XA, Hudes ES, Johnson MO, Ruel T, Neilands TB. A Mobile Health App (WYZ) for Engagement in Care and Antiretroviral Therapy Adherence Among Youth and Young Adults Living With HIV: Single-Arm Pilot Intervention Study. JMIR Form Res. 2021 Aug 31;5(8):e26861. doi: 10.2196/26861. PMID 34463622
- [Result] Lisha NE, Neilands TB, Erguera XA, Saberi P. Development of the Mobile Technology Vulnerability Scale among Youth and Young Adults Living with HIV. Int J Environ Res Public Health. 2021 Apr 15;18(8):4170. doi: 10.3390/ijerph18084170. PMID 33920803

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Intervention
Started | 79
Completed | 69
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1: Intervention
Number analyzed (Participants) | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 79
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 declined to answer
  Participants
    number analyzed (Participants) | 78
    Female | 9
    Male | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 20
  White | 18
  More than one race | 21
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 79

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Rate of Participant Recruitment
Description: Recruit at least 55 participants (i.e. 70% of target N)
Time Frame: 8 Months
Population: Overall Number of Participants Analyzed represents number of participants screened for study interest prior to recruitment/enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Intervention
Number analyzed (Participants) | 92
Participants | 79

2. Primary Outcome: Feasibility: Frequency of WYZ Access
Description: Mean number of logins/week over the 6 month period of using WYZ
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: Mean logins/week
Arm/Group | Arm 1: Intervention
Number analyzed (Participants) | 79
Mean logins/week | 5.3 (5.6)

3. Primary Outcome: Feasibility: Length of Session (Minutes)
Description: Mean minutes/week spent in the app over the 6 month period of using WYZ
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: Mean minutes/week
Arm/Group | Arm 1: Intervention
Number analyzed (Participants) | 79
Mean minutes/week | 8.7 (5)

4. Primary Outcome: Feasibility: Rate of Use of ART Adherence Tracking
Description: Mean percentage of times/week that participants tracked ART adherence in the app over 6 months of using WYZ. E.g. 3 mean times/week = 43% mean/week.
Time Frame: 6 Months
Measure: Mean (Full Range); unit: % mean times tracked/week
Arm/Group | Arm 1: Intervention
Number analyzed (Participants) | 79
% mean times tracked/week | 58 [0 to 100]

5. Primary Outcome: Feasibility: Rate of Communication With Peers
Description: Mean number of postings of chat topics on the My Community chat per person per week, over 6 months of using WYZ
Time Frame: 6 Months
Measure: Mean (Full Range); unit: Mean postings/person/week
Arm/Group | Arm 1: Intervention
Number analyzed (Participants) | 79
Mean postings/person/week | 4.8 [1 to 42]

6. Secondary Outcome: Acceptability: Participant Retention
Description: Percentage of individuals who enrolled and completed the study at 6 months
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Intervention
Number analyzed (Participants) | 79
Participants | 69

7. Secondary Outcome: Acceptability: Overall App Experience
Description: Percent of participants who rated their overall experience with the app as excellent to very good
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Intervention
Number analyzed (Participants) | 69
Participants | 53

8. Secondary Outcome: Acceptability: Privacy, Security, and Anonymity
Description: Percent of participants who reported being extremely to somewhat comfortable with the security, privacy, and anonymity of WYZ
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Intervention
Number analyzed (Participants) | 69
Participants | 69

9. Secondary Outcome: Acceptability: Continue Using WYZ
Description: Percent of participants who stated that they would be extremely to somewhat likely to continue to use WYZ
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Intervention
Number analyzed (Participants) | 69
Participants | 57

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Arm 1: Intervention
All-Cause Mortality (participants affected / at risk) | 0/79
Serious Adverse Events (participants affected / at risk) | 0/79
Other Adverse Events (participants affected / at risk) | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT03587857/Prot_SAP_000.pdf